CLINICAL TRIAL: NCT05445232
Title: A Multiple-Dose Drug-Drug Interaction Study to Determine the Effect of LY3437943 on Drug Metabolizing Enzymes
Brief Title: A Drug-Drug Interaction (DDI) Study of LY3437943 in Obese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 18476; J1I-MC-GZBI (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04-01

CONDITIONS: Obesity
Keywords: Overweight; Obesity; Drug Interaction; Cocktail; Pharmacokinetic
MeSH Terms: conditions — Obesity; Overweight | interventions — retatrutide; Midazolam; Warfarin; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY3437943 + Drug Cocktail (Experimental): Midazolam in combination with warfarin and caffeine (drug cocktail) administered orally followed by LY3437943 administered subcutaneously (SC) in week 1.
  At weeks 8, 12, & 16, the LY3437943 will be administered SC on Day 1 followed by midazolam in combination with warfarin and caffeine (drug cocktail) administered orally on Day 2.
  Interventions: Drug: LY3437943; Drug: Midazolam; Drug: Warfarin; Drug: Caffeine

INTERVENTIONS:
Drug: LY3437943 — Administered SC.
Drug: Midazolam — Administered orally.
Drug: Warfarin — Administered orally.
Drug: Caffeine — Administered orally.

SUMMARY:
The main purpose of this study is to determine the effect of LY3437943 when administered subcutaneously on the levels of midazolam, warfarin and caffeine in the blood stream when administered orally as a drug cocktail in obese participants. This study will last up to approximately 25 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) within the range 27.0 to 40.0 kilograms per meter squared (kg/m²)
* Male and female participants of childbearing potential who agree to use contraceptive methods

Exclusion Criteria:

* Have a history of diabetes or current diagnosis of diabetes
* History or presence of a of significant bleeding disorder
* Participants with significant comorbidity
* Participants receiving treatment with midazolam, warfarin, inhibitors or inducers of cytochrome P450 (CYP) -1A2, CYP2C9, or CYP3A4 enzymes, or drugs are CYP substrates and have a narrow therapeutic index

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Midazolam | Predose up to 24 hours postdose
  PK: AUC[0-∞] of Midazolam
PK: Maximum Observed Concentration (Cmax) of Midazolam | Predose up to 24 hours postdose
  PK: Cmax of Midazolam
PK: AUC[0-∞] of Warfarin | Predose up to 96 hours postdose
  PK: AUC[0-∞] of Warfarin
PK: Cmax of Warfarin | Predose up to 96 hours postdose
  PK: Cmax of Warfarin
PK: AUC[0-∞] of Caffeine | Predose up to 48 hours postdose
  PK: AUC[0-∞] of Caffeine
PK: Cmax of Caffeine | Predose up to 48 hours postdose
  PK: Cmax of Caffeine

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Covance Clinical Research Unit, Daytona Beach, Florida
  - Covance Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No